CLINICAL TRIAL: NCT03382561
Title: Randomized Phase II Clinical Trial of Cisplatin/Carboplatin and Etoposide (CE) Alone or in Combination With Nivolumab as Frontline Therapy for Extensive Stage Small Cell Lung Cancer (ED-SCLC)
Brief Title: Cisplatin/Carboplatin and Etoposide With or Without Nivolumab in Treating Patients With Extensive Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-02367; NCI-2017-02367 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA5161 (Other: ECOG-ACRIN Cancer Research Group); EA5161 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2017-12-21; First posted 2017-12-26 (Actual); Results first posted 2023-06-23 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Extensive Stage Lung Small Cell Carcinoma; Recurrent Lung Small Cell Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Etoposide; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (nivolumab, CE) (Experimental): Patients receive nivolumab IV over 30 minutes on day 1, carboplatin IV over 30-60 minutes on day 1 or cisplatin IV over 60-120 minutes on day 1, and etoposide IV over 60-120 minutes on days 1-3. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients continue to receive nivolumab IV over 30 minutes every 2 weeks for up to 2 years.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Etoposide; Biological: Nivolumab
- Arm B (CE) (Active Comparator): Patients receive carboplatin IV over 30-60 minutes on day 1 or cisplatin IV over 60-120 minutes on day 1, and etoposide IV over 60-120 minutes on days 1-3. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
  Arms: Arm A (nivolumab, CE)

SUMMARY:
This randomized phase II clinical trial studies whether the addition of nivolumab to cisplatin (or carboplatin) and etoposide will improve outcomes when treating patients with extensive stage small cell lung cancer. Chemotherapy drugs, such as cisplatin, carboplatin, and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving cisplatin/carboplatin and etoposide together with nivolumab may work better in treating patients with extensive stage small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the progression-free survival (PFS) of patients with extensive stage small cell lung cancer (ED-SCLC) treated with cisplatin/carboplatin and etoposide (CE) or CE with nivolumab (CEN) as front-line treatment.

SECONDARY OBJECTIVES:

I. To estimate overall survival of patients with ED-SCLC treated with cisplatin/carboplatin and etoposide (CE) or CE with nivolumab (CEN) as front-line treatment.

II. To assess best overall response rate after treatment with CE with or without nivolumab as first line treatment.

III. To evaluate the toxicity profile of nivolumab with CE.

EXPLORATORY OBJECTIVES:

I. To evaluate immune biomarkers and biomarkers correlatives. II. To evaluate serial circulating tumor deoxyribonucleic acid (DNA) and explore whether clinical outcome is associated with fluctuations in DNA levels following the administration of therapy.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive nivolumab intravenously (IV) over 30 minutes on day 1, carboplatin IV over 30-60 minutes on day 1 or cisplatin IV over 60-120 minutes on day 1, and etoposide IV over 60-120 minutes on days 1-3. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients continue to receive nivolumab IV over 30 minutes every 2 weeks for up to 2 years.

ARM B: Patients receive carboplatin IV over 30-60 minutes on day 1 or cisplatin IV over 60-120 minutes on day 1, and etoposide IV over 60-120 minutes on days 1-3. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months if the patient is less than 2 years from registration, every 6 months if the patient is 2-3 years from registration, and yearly for up to 5 years from study enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed extensive stage small cell lung cancer and must be a candidate for systemic therapy; NOTE: The extensive disease SCLC classification for this protocol includes all patients with disease sites not defined as limited stage; limited stage disease category includes patients with disease restricted to one hemithorax with regional lymph node metastases, including hilar, ipsilateral and contralateral mediastinal, and/or ipsilateral supraclavicular nodes; extensive disease patients are defined as those patients with extrathoracic metastatic disease, malignant pleural effusion, bilateral or contralateral supraclavicular adenopathy; patients with locally recurrent SCLC who are not eligible for curative intent chemoradiation are eligible
* Patients must have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Absolute neutrophil count >= 1,500/mm^3 (must be obtained =< 7 days prior to protocol registration)
* Platelets >= 100,000/mm^3 (must be obtained =< 7 days prior to protocol registration)
* Leukocytes >= 3000/mm^3 (must be obtained =< 7 days prior to protocol registration)
* Hemoglobin >= 9 g/dL (must be obtained =< 7 days prior to protocol registration)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (except subjects with Gilbert syndrome, who can have total bilirubin < 3 mg/dL) (must be obtained =< 7 days prior to protocol registration)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 3 X institutional upper limit of normal (ULN) (=< 5 X if liver function test [LFT] elevations due to known liver metastases) (must be obtained =< 7 days prior to protocol registration)
* Serum creatinine =< 1.5 x ULN or calculated creatinine clearance > 50 mL/min (using the Cockcroft-Gault formula) (must be obtained =< 7 days prior to protocol registration)
* Patients are eligible if central nervous system (CNS) metastases are adequately treated and neurological symptoms have returned to baseline or are controlled for at least 2 weeks prior to enrollment; in addition, subjects must be either off corticosteroids, or on a stable or decreasing dose of =< 10 mg daily prednisone (or equivalent); patients with untreated CNS metastases are eligible if they are not symptomatic and the lesions are less than 1 cm in size
* Patients cannot have had prior chemotherapy or biologic therapy for extensive stage small cell lung cancer for front line treatment; patients receiving prior whole brain radiation cannot register within 7 days after completion of radiation, and must have resolved adverse events attributed to radiation to =< grade 1; a 1-week washout is permitted for palliative radiation (=< 2 weeks of radiotherapy) to non-CNS disease
* Patients who have received prior chemoradiation treatment with chemotherapy regimen including cisplatin or carboplatin/etoposide for limited-stage SCLC are eligible if treated with curative intent at least 6 months since last treatment from diagnosis of extensive-stage SCLC
* Patients may not be receiving any other investigational agents while on study
* Women of childbearing potential (WOCBP) and males who are sexually active with WOCBP must use an accepted and effective method of contraception or abstain from sexual intercourse for at least one week prior to the start of treatment, and continue for 5 months after the last dose of protocol treatment for women of childbearing potential and 7 months after the last dose of protocol treatment for males who are sexually active with WOCBP
* No prior or current invasive malignancy (except non-melanomatous skin cancer, localized bladder and prostate cancer) unless disease free for a minimum of 2 years (for example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible);
* No prior systemic treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways;
* No patients with an active, known or suspected autoimmune disease and neuromuscular paraneoplastic syndromes including but not limited to myasthenia gravis, Lambert-Eaton myasthenic syndrome, limbic encephalitis, myositis, Guillain-Barre; subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* No patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 7 days of randomization; inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease
* No patients with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity
* No history of severe hypersensitivity reaction to any monoclonal antibody or allergy to study drug components

Exclusion Criteria:

* Patients must not have history of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab or other agents used in the study
* Women must not be pregnant or breast-feeding; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the agents used in this study, breastfeeding must be discontinued or the subject is not eligible for the study; all females of childbearing potential must have a blood test or urine study, with a minimum sensitivity 50 mlU/L or equivalent units of human chorionic gonadotropin (HCG), within 14 days prior to registration to rule out pregnancy; a female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e. has had menses at any time in the preceding 24 consecutive months)
* Patient must not have leptomeningeal disease
* Patients must NOT have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Any positive test for hepatitis B virus or hepatitis C virus indicating acute or chronic infection, patients are excluded
* Patients are ineligible if they received a live, attenuated vaccine within 4 weeks before randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2025-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ticiana A Leal, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (779):
- United States (779):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Northbay Cancer Center, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Good Samaritan Hospital - Cancer Centers of Colorado, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner McKee Medical Center, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Middlesex Hospital, Middletown, Connecticut
  - Veterans Affairs Connecticut Healthcare System-West Haven Campus, West Haven, Connecticut
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Bayhealth Hospital Sussex Campus, Milford, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - The Watson Clinic, Lakeland, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Low Country Cancer Care, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Summit Cancer Care-Candler, Savannah, Georgia
  - Lewis Hall Singletary Oncology Center, Thomasville, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Freeport Memorial Hospital/Leonard C Ferguson Cancer Center, Freeport, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - North Shore Medical Center, Skokie, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Coffeyville Regional Medical Center, Coffeyville, Kansas
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Baptist Health Corbin, Corbin, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Elizabeth Healthcare Edgewood, Edgewood, Kentucky
  - Saint Elizabeth Healthcare Fort Thomas, Fort Thomas, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Oncology Center of The South Incorporated, Houma, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - MaineHealth Waldo Hospital, Belfast, Maine
  - MaineHealth Maine Medical Center - Biddeford, Biddeford, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth Cancer Care and IV Therapy - Sanford, Sanford, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - UPMC Western Maryland, Cumberland, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Simonds-Sinon Regional Cancer Center, Fitchburg, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Mercy Medical Center, Springfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Beth Israel Deaconess Medical Center/Winchester Center for Cancer Care, Winchester, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - McLaren Cancer Institute-Bloomfield, Bloomfield, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Ascension Borgess Hospital, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Hattiesburg Clinic - Hematology/Oncology Clinic, Hattiesburg, Mississippi
  - Forrest General Hospital / Cancer Center, Hattiesburg, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Faith Regional Health Services Carson Cancer Center, Norfolk, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Nebraska Cancer Specialists - Omaha, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Oncology Hematology West PC, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Regional West Medical Center Cancer Center, Scottsbluff, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - GenesisCare USA - Henderson, Henderson, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - GenesisCare USA - Las Vegas, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - GenesisCare USA - Vegas Tenaya, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - GenesisCare USA - Fort Apache, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Ocean University Medical Center, Brick, New Jersey
  - Bayshore Community Hospital, Holmdel, New Jersey
  - Meridian Health Village at Jackson, Jackson, New Jersey
  - Southern Ocean County Medical Center, Manahawkin, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Inspira Medical Center Mullica Hill, Mullica Hill, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Neurosurgeons of New Jersey-Ridgewood, Ridgewood, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Valley Medical Group - Wayne Multispecialty Practice, Wayne, New Jersey
  - Valley Health System-Hematology/Oncology, Westwood, New Jersey
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Garnet Health Medical Center, Middletown, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - SUNY Upstate Medical Center-Community Campus, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospital, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Bristol Regional Medical Center, Bristol, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Johnson City, Johnson City, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Ballad Health Cancer Care - Bristol, Bristol, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Augusta Health Center for Cancer and Blood Disorders, Fishersville, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours DePaul Medical Center, Norfolk, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Bon Secours Health Center at Harbour View, Suffolk, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Wu J, Zhang A, Li L, Liu S, Yang F, Yang R. Meta-analysis of the Efficacy and Tolerability of Immune Checkpoint Inhibitors Combined With Chemotherapy in First-line Treatment of Small Cell Lung Cancer. Clin Ther. 2021 Mar;43(3):582-593.e2. doi: 10.1016/j.clinthera.2020.12.017. Epub 2021 Jan 25. PMID 33509647

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study activated on May 2, 2018, and closed to accrual on December 7, 2018 after enrolling a total of 160 patients.
Groups:
- Arm A (Cisplatin/Carboplatin, Etoposide and Nivolumab; CEN): Patients receive nivolumab IV at 360 mg over 30 minutes on day 1, carboplatin AUC 5 or 6 IV over 30-60 minutes on day 1 or cisplatin at 75 mg/m2 IV over 60-120 minutes on day 1, and etoposide at 100 mg/m2 IV over 60-120 minutes on days 1-3. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients continue to receive nivolumab IV over 30 minutes every 2 weeks for up to 2 years.
- Arm B (Cisplatin/Carboplatin and Etoposide; CE): Patients receive carboplatin AUC 5 or 6 IV over 30-60 minutes on day 1 or cisplatin at 75 mg/m2 IV over 60-120 minutes on day 1, and etoposide at 100 mg/m2 IV over 60-120 minutes on days 1-3. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm A (Cisplatin/Carboplatin, Etoposide and Nivolumab; CEN) | Arm B (Cisplatin/Carboplatin and Etoposide; CE)
Started | 80 | 80
Received Treatment | 77 | 74
Eligible and Treated Patients | 75 | 69
Completed | 4 | 47
Not Completed | 76 | 33
Not completed — Disease progression | 47 | 6
Not completed — Adverse Event | 10 | 2
Not completed — Death | 8 | 3
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Alternative therapy | 2 | 8
Not completed — Never started treatment | 3 | 6
Not completed — Lack of Efficacy | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Other complicating disease | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Cisplatin/Carboplatin, Etoposide and Nivolumab; CEN) | Arm B (Cisplatin/Carboplatin and Etoposide; CE) | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Continuous [Median (Full Range); unit: years] | 64 [44 to 85] | 65 [43 to 86] | 65 [43 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 44 | 89
  Male | 35 | 36 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 78 | 78 | 156
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 0 | 7
  White | 73 | 76 | 149
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from randomization to documented disease progression or death from any cause, whichever occurs first. Patients who have not experienced an event of interest by the time of analysis will be censored at the date they are last known to be alive and progression-free.
  Progression was evaluated using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Progression was defined as appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions, or at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Every 6 weeks for 6 months, then every 8 weeks until 1 year, and then every 12 weeks until being off treatment or end of observation. Thereafter every 3 months if < 2 years from registration, every 6 months for years 2-3, and yearly up to 3 years 9 months
Population: Eligible and treated patients were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Cisplatin/Carboplatin, Etoposide and Nivolumab; CEN) | Arm B (Cisplatin/Carboplatin and Etoposide; CE)
Number analyzed (Participants) | 75 | 69
months | 5.5 [4.3 to 5.9] | 4.9 [4.5 to 5.7]
Statistical Analysis 1: Comparison: Arm A (Cisplatin/Carboplatin, Etoposide and Nivolumab; CEN) vs Arm B (Cisplatin/Carboplatin and Etoposide; CE); Test type: Superiority; p = 0.17, Log Rank; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.55 to 1.11] — Hazard ratio: Arm A (CEN)/Arm B (CE)

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from maintenance randomization until death of any cause.
Time Frame: Every 6 weeks for 6 months, then every 8 weeks until 1 year, and then every 12 weeks until off treatment or end of observation. Then every 3 months if < 2 years from registration, every 6 months for years 2-3, and yearly up to 3 years 9 months.
Population: Eligible and treated patients were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Cisplatin/Carboplatin, Etoposide and Nivolumab; CEN) | Arm B (Cisplatin/Carboplatin and Etoposide; CE)
Number analyzed (Participants) | 75 | 69
months | 11.2 [8.8 to 14.2] | 8.1 [7.2 to 9.6]

3. Secondary Outcome: Response Rate
Description: Best overall response was evaluated using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Response was defined as complete response (CR) or partial response (PR).
  CR: Disappearance of all lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: as for outcome 1
Population: Eligible and treated patients were included in this analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Cisplatin/Carboplatin, Etoposide and Nivolumab; CEN) | Arm B (Cisplatin/Carboplatin and Etoposide; CE)
Number analyzed (Participants) | 75 | 69
proportion of participants | 0.77 [0.66 to 0.86] | 0.80 [0.68 to 0.88]

4. Other Pre Specified Outcome: PD-L1 Expression Level
Time Frame: Assessed at baseline and 6 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Association Between Circulating Tumor DNA and Clinical Outcome
Time Frame: circulating tumor DNA was assessed at baseline and 6 weeks; clinical outcomes were assessed every 3 months for patients < 2 years from registration, every 6 months if patient is 2-3 years from registration, and annually until 5 years from registration
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed every 6 weeks while on treatment and for 30 days after the end of treatment for adverse events. All-cause mortality was assessed up to 4 years.
Description: All patients were included in the all-cause mortality analysis. Only patients who received treatment were included in the analysis of adverse events.
Arm/Group | Arm A (Cisplatin/Carboplatin, Etoposide and Nivolumab; CEN) | Arm B (Cisplatin/Carboplatin and Etoposide; CE)
All-Cause Mortality (participants affected / at risk) | 67/80 | 74/80
Serious Adverse Events (participants affected / at risk) | 59/77 | 49/74
Other Adverse Events (participants affected / at risk) | 76/77 | 73/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Cisplatin/Carboplatin, Etoposide and Nivolumab; CEN) (N=77) | Arm B (Cisplatin/Carboplatin and Etoposide; CE) (N=74)
Hearing impaired (Ear and labyrinth disorders) | 1 | 1
Anemia (Blood and lymphatic system disorders) | 17 | 11
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 3
Atrial fibrillation (Cardiac disorders) | 1 | 1
Fatigue (General disorders) | 10 | 5
Infusion related reaction (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0
Endocrine disorders - Other, specify (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0
Anaphylaxis (Immune system disorders) | 1 | 0
Immune system disorders - Other, specify (Immune system disorders) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 4 | 1
Sepsis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Alkaline phosphatase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 13 | 13
Neutrophil count decreased (Investigations) | 36 | 38
Platelet count decreased (Investigations) | 14 | 12
Serum amylase increased (Investigations) | 1 | 0
Weight loss (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 13 | 16
Investigations - Other, specify (Investigations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 4 | 0
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 1
Hallucinations (Psychiatric disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 2
Thromboembolic event (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Cisplatin/Carboplatin, Etoposide and Nivolumab; CEN) (N=77) | Arm B (Cisplatin/Carboplatin and Etoposide; CE) (N=74)
Anemia (Blood and lymphatic system disorders) | 59 | 57
Edema limbs (General disorders) | 5 | 3
Fatigue (General disorders) | 53 | 55
Fever (General disorders) | 6 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 25 | 28
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 18 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13 | 1
Hyperthyroidism (Endocrine disorders) | 4 | 0
Hypothyroidism (Endocrine disorders) | 9 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 4
Constipation (Gastrointestinal disorders) | 9 | 9
Diarrhea (Gastrointestinal disorders) | 23 | 12
Dry mouth (Gastrointestinal disorders) | 7 | 8
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 | 4
Mucositis oral (Gastrointestinal disorders) | 5 | 4
Nausea (Gastrointestinal disorders) | 39 | 34
Vomiting (Gastrointestinal disorders) | 8 | 6
Alanine aminotransferase increased (Investigations) | 7 | 8
Alkaline phosphatase increased (Investigations) | 14 | 2
Aspartate aminotransferase increased (Investigations) | 12 | 9
Creatinine increased (Renal and urinary disorders) | 12 | 11
Lymphocyte count decreased (Investigations) | 30 | 20
Neutrophil count decreased (Investigations) | 24 | 23
Platelet count decreased (Investigations) | 27 | 30
Weight loss (Investigations) | 12 | 6
White blood cell decreased (Investigations) | 25 | 17
Investigations - Other, specify (Investigations) | 4 | 5
Anorexia (Metabolism and nutrition disorders) | 31 | 26
Dehydration (Metabolism and nutrition disorders) | 1 | 5
Hyperglycemia (Metabolism and nutrition disorders) | 7 | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 | 11
Hypocalcemia (Metabolism and nutrition disorders) | 6 | 3
Hypokalemia (Metabolism and nutrition disorders) | 9 | 12
Hypomagnesemia (Metabolism and nutrition disorders) | 7 | 10
Hyponatremia (Metabolism and nutrition disorders) | 9 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 5
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 8 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Dizziness (Nervous system disorders) | 12 | 6
Dysgeusia (Nervous system disorders) | 11 | 9
Headache (Nervous system disorders) | 4 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 9 | 8
Insomnia (Psychiatric disorders) | 6 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Proteinuria (Renal and urinary disorders) | 4 | 2
Hypotension (Vascular disorders) | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/61/NCT03382561/Prot_SAP_000.pdf